CLINICAL TRIAL: NCT02303327
Title: Phase III Study of Hypofractionated, Dose Escalation Radiotherapy Vs. Conventional Pelvic Radiation Therapy Followed by HDR Brachy Boost for High Risk Adenocarcinoma of the Prostate (PCS-VI)
Brief Title: Comparative Study of Radiotherapy Treatments to Treat High Risk Prostate Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Radiation Oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS VI
Record Dates: First submitted 2014-11-10; First posted 2014-11-27 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADT+EBRT+ HDR brachytherapy boost (Other): Standard fractionation radiotherapy: 46 Gy in 23 fractions (EBRT) and a 15-Gy HDRB boost in conjunction with 28 months of androgen deprivation therapy (ADT).
  Interventions: Radiation: EBRT + HDR brachytherapy boost; Drug: Androgen deprivation therapy
- ADT+Hypofractionated Dose Escalation RT (Active Comparator): Hypofractionated dose escalation radiotherapy: 68 Gy in 25 fractions in conjunction with 28 months of androgen deprivation therapy (ADT).
  Interventions: Radiation: Hypofractionated Dose Escalation Radiotherapy; Drug: Androgen deprivation therapy

INTERVENTIONS:
Radiation: EBRT + HDR brachytherapy boost — Standard radiotherapy (EBRT, 23 fractions) with the addition of High Dose-Rate (HDR) brachytherapy boost within 3 weeks of beginning or finishing the EBRT.
  Arms: ADT+EBRT+ HDR brachytherapy boost
Radiation: Hypofractionated Dose Escalation Radiotherapy — Radiation therapy (higher radiation dose per treatment) will be given once a day, five days a week, over approximately 5 weeks.
  Arms: ADT+Hypofractionated Dose Escalation RT
Drug: Androgen deprivation therapy — 28 months of androgen deprivation therapy (injections every 4 months for a total of 28 months)
  Other Names: ADT

SUMMARY:
In North America, the number of new cases of prostate cancer increases every year. Many efforts have been made to develop more efficient and safer curative treatments for high risk prostate cancer patients.

This phase III clinical trial is designed to compare the safety of a standard pelvic external beam radiation therapy (EBRT) combined with a high dose rate brachytherapy (HDRB) boost (direct insertion of radiation source over a period of minutes via flexible needles temporarily inserted in the prostate) to a shorter course of hypofractionated dose escalation radiotherapy (larger radiation dose per daily treatment) in patients with high risk prostate cancer.

The investigators plan to recruit 296 patients across Quebec who will be randomized in either treatment plan.

DETAILED DESCRIPTION:
In North America, the number of new cases of prostate cancer increases every year. To this day, the standard curative treatment for high risk prostate cancer patients is external beam radiation therapy (EBRT) combined with hormonal manipulation (Luteinizing hormone-releasing hormone LHRH agonists such as Eligard) to lower levels of testosterone to slow down or even stop the growth of prostate cancer. It has been recently demonstrated that combination of high dose rate brachytherapy (HDRB) boost (direct insertion of radiation source in the prostate for killing the tumor) to EBRT could be an effective treatment for prostate cancer patients. On the other hand, other recent studies have suggested that dose escalation and hypofractionated radiation delivery (larger radiation dose per daily treatment) can be more efficient than standard fractionation in prostate cancer patients.

This phase III clinical trial is designed to compare the safety of a conventional pelvic EBRT combined with a HDRB boost (i.e. 46 Gy in 23 fractions followed by a 15-Gy HDRB boost) to a shorter course of hypofractionated dose escalation radiotherapy (i.e. 68 Gy in 25 fractions) in patients with high risk prostate cancer. The patients will be randomized to either of the two different courses of treatment. All the patients will be also treated with hormonal therapy for a total duration of 28 months (2 months before radiation therapy (RT), 2 months during RT and for 24 months after RT). The patients will undergo different test before the treatment, such as bone scan, blood test, CT scan and bone density. The patient's follow-up will be the first month after start of RT, every 4 months for the first 2 years, then every 6 months the third year and then annually for 10 years. On every visit, the patient will undergo digital rectal examination (DRE) as well as evaluation of testosterone and prostate specific antigen (PSA) levels.

The safety of the new course of radiation therapy will be evaluated by the acute (at and before 90 days) and delayed toxicities (at 90 days, at 180 days and after) measured by Common Terminology Criteria for Adverse Events (CTCAE version 4). We will also determine Biochemical Failure Free Survival, Distant Metastasis Free Survival, Disease Specific Survival, Overall Survival and the Health-related Quality of Life using the Expanded Prostate Cancer Index Composite (EPIC). We will also monitor the development of gastrointestinal and genitourinary toxicities and establish the predictive value of PTEN deletion and TMPRSS2ETS fusion (genetic markers to predict the nature and progression of prostate tumors).

This study will be conducted through the Genitourinary Radiation Oncology Group of Quebec (GROUQ) in 12 selected radiation oncology centers. We plan to recruit 296 patients across Quebec and the recruitment should be completed within 24 months of activation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within 6 months prior to randomization, (if longer than 6 months, needs to be approved by the PI).
* Clinical stage including at least one of the following: T3 or T4, Gleason Score > 8, and/ or Prostate-specific antigen (PSA) > 20 (ng/ml or μg/L).
* Pelvic and para-aortic lymph nodes must be negative on CT scan or MRI of the abdomen and pelvis performed within 12 (recommended time limit, may exceed in certain cases) weeks prior to randomization. For patients who have started androgen suppression prior to randomization, CT or MRI may be done after start of therapy, provided it is done no more than 28 days following start of androgen suppression therapy (any lymph node appearing > 1.5 cm on CT or MRI must be histologically negative by either needle aspirate or lymph node dissection performed within 12 weeks prior to randomization).
* Investigations, including chest x-ray (CXR is recommended and not mandatory) CT scan and bone scan (with radiographs of suspicious areas) have been performed within 12 weeks (recommended time limit) prior to randomization and are negative for metastases. For patients who have started androgen suppression prior to randomization, bone scan may be done up to and including 28 days after the commencement of therapy.
* Patients will have had a PSA test done at the time of diagnosis. This PSA test could be repeated within 28 days prior to randomization. The PSA value used to confirm high risk disease and the value to be entered on the eligibility checklist must be the higher of these two values. These criteria will be the same regardless of whether or not the patient has initiated hormone therapy prior to randomization.
* The patient may have received prior androgen suppression therapy provided that androgen suppression therapy commenced no more than 28 days prior to randomization.
* The patient must not have received any cytotoxic anticancer therapy for prostate cancer prior to randomization. Patients may have received treatment with a 5-alpha-reductase inhibitor (e.g. Finasteride) for benign prostatic hypertrophy (BPH), which must have been discontinued prior to the randomization.
* ECOG performance status must be 0 or 1.
* Hematology and Biochemistry: Laboratory requirements have been done within 28-42 days prior to randomization: hemoglobin > 100 g/L, absolute Neutrophils > 1.5 x 109/L, platelets > 100 x 109/L, serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Patients with a history of other malignancies, except: non-melanoma skin cancer; or other solid tumours curatively treated with no evidence of disease for > 5 years.
* The presence of small-cell or transitional-cell carcinoma in the biopsy specimen.
* Patients who had previous chemotherapy for carcinoma of the prostate.
* Patients who had prior surgical treatment for carcinoma of the prostate apart from trans-urethral resection, including bilateral orchiectomy.
* Patients with any contraindication to pelvic radiotherapy: including, but not limited to, previous pelvic radiotherapy. Inflammatory bowel disease (at the discretion of the treating oncologist) or severe bladder irritability.
* Patients with serious non malignant disease resulting in a life expectancy less than 3 years.
* Other serious illness, psychiatric or medical condition that would not permit the patient to be managed according to the protocol including active uncontrolled infection and significant cardiac dysfunction. Patients with medical conditions that would contraindicate the treatment regimen outlined in the protocol [e.g. intake of study drugs].
* Known hypersensitivity to any protocol-indicated study medications.
* Presence of bilateral hip replacement prostheses.
* Patients with history of severe congestive heart failure will not be eligible.
* Patients with congenital long QT syndrome or patients taking Class IA, Class III or Class IC anti-arrhythmic medications will require a cardiologist's evaluation prior to eligibility assessment. Patients with cardiovascular diseases can be included as long as the benefits of androgen deprivation therapy outweigh the potential risk of cardiovascular events.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-01; Primary Completion 2026-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Acute and delayed toxicity differences measured by Common Terminology Criteria for Adverse Events (CTCAE) version 4. | The acute toxicity will be evaluated at or before 90 days and for the delayed toxicity, it will be determined at 90 -180 days and after (persisting or appearing after 180 days).

SECONDARY OUTCOMES:
Freedom from biochemical failure measured by PSA level. | At 3 and 5 years.
  an increase by 2 ng/mL or more above the nadir PSA is considered as biochemical failure
Rate of local failures measured by number of recurrences in the prostate. | At 3 and 5 years.
Rate of regional failures measured by number of recurrences in the lymph nodes. | At 3 and 5 years.
Rate of distant failures measured by number of metastases. | At 3 and 5 years.
Disease specific survival measured by number of deaths associated to the prostate cancer. | At 5 years.
Disease overall survival measured by the number of deaths after 5 years. | At 5 years.
Health-related quality of life measured by using Expanded Prostate Cancer Index Composite (EPIC) questionnaire | At every routine visit (baseline, 3 to 4 weeks after RT, every 4 months for 2 years, every 6 months the 3 following years and then annually until 10 years).
Correlation of dose-volume histogram of the rectum and bladder by studying wall and whole organ volumes to the development of gastrointestinal (GI) and genitourinary (GU) toxicity. | At 180 days post treatment
Predictive value of the PTEN deletion and TMPRSS2-ETS gene fusion in high risk prostate cancer patients. | At the time when biopsy is done, < 6 months before randomization of participant
  looking for correlation between these known gene mutations and local and/or distal recurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital, McGill University
Locations (12):
- Canada (12):
  - Eastern Health, St. John's, Newfoundland and Labrador
  - Lawson Health Research Institute, London, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre Hospitalier des Vallées de l'Outaouais, Hôpital de Gatineau, Gatineau, Quebec
  - CHUM Notre-Dame, Montreal, Quebec
  - Montréal General Hospital, Montreal, Quebec
  - Jewish General Hospital, McGill University, Montreal, Quebec
  - CHUQ, L'Hôtel-Dieu de Québec, Québec, Quebec
  - Centre de santé Rimouski-Neigette, Rimouski, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
  - Centre Hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Background] Canadian Cancer Statistics 2010. www.cancer.ca.
- [Background] Levy IG, Gibbons L, Collins JP, Perkins DG, Mao Y. Prostate cancer trends in Canada: rising incidence or increased detection? CMAJ. 1993 Sep 1;149(5):617-24. PMID 8364818
- [Background] Pilepich MV, Winter K, John MJ, Mesic JB, Sause W, Rubin P, Lawton C, Machtay M, Grignon D. Phase III radiation therapy oncology group (RTOG) trial 86-10 of androgen deprivation adjuvant to definitive radiotherapy in locally advanced carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1243-52. doi: 10.1016/s0360-3016(01)01579-6. PMID 11483335
- [Background] McCammon R, Rusthoven KE, Kavanagh B, Newell S, Newman F, Raben D. Toxicity assessment of pelvic intensity-modulated radiotherapy with hypofractionated simultaneous integrated boost to prostate for intermediate- and high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):413-20. doi: 10.1016/j.ijrobp.2008.10.050. Epub 2009 Apr 11. PMID 19362783
- [Background] Pervez N, Small C, MacKenzie M, Yee D, Parliament M, Ghosh S, Mihai A, Amanie J, Murtha A, Field C, Murray D, Fallone G, Pearcey R. Acute toxicity in high-risk prostate cancer patients treated with androgen suppression and hypofractionated intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):57-64. doi: 10.1016/j.ijrobp.2009.01.048. PMID 19395192
- [Background] Hong TS, Tome WA, Jaradat H, Raisbeck BM, Ritter MA. Pelvic nodal dose escalation with prostate hypofractionation using conformal avoidance defined (H-CAD) intensity modulated radiation therapy. Acta Oncol. 2006;45(6):717-27. doi: 10.1080/02841860600781781. PMID 16938815
- [Background] Arcangeli G, Saracino B, Gomellini S, Petrongari MG, Arcangeli S, Sentinelli S, Marzi S, Landoni V, Fowler J, Strigari L. A prospective phase III randomized trial of hypofractionation versus conventional fractionation in patients with high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):11-8. doi: 10.1016/j.ijrobp.2009.07.1691. Epub 2010 Jan 4. PMID 20047800
- [Background] Hsu IC, Pickett B, Shinohara K, Krieg R, Roach M 3rd, Phillips T. Normal tissue dosimetric comparison between HDR prostate implant boost and conformal external beam radiotherapy boost: potential for dose escalation. Int J Radiat Oncol Biol Phys. 2000 Mar 1;46(4):851-8. doi: 10.1016/s0360-3016(99)00501-5. PMID 10705005
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316
- [Background] Guix B, et al. Treatment of Intermediate-or High-risk Prostate Cancer by Dose Escalation with High-dose 3D-conformal Radiotherapy (HD-3D-CRT) or Low-dose 3D-conformal Radiotherapy Plus HDR Brachytherapy (LD-3D-CRT+HDR-B): Early Results of a Prospective Comparative Trial. Int J Radiat Oncol Biol Phys. 78[3], S78. 11-1-2010.
- [Background] Cury FL, Duclos M, Aprikian A, Patrocinio H, Kassouf W, Shenouda G, Faria S, David M, Souhami L. Single-fraction high-dose-rate brachytherapy and hypofractionated external beam radiation therapy in the treatment of intermediate-risk prostate cancer - long term results. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1417-23. doi: 10.1016/j.ijrobp.2011.05.025. Epub 2011 Jul 23. PMID 21784585
- [Background] Roach M 3rd, Bae K, Speight J, Wolkov HB, Rubin P, Lee RJ, Lawton C, Valicenti R, Grignon D, Pilepich MV. Short-term neoadjuvant androgen deprivation therapy and external-beam radiotherapy for locally advanced prostate cancer: long-term results of RTOG 8610. J Clin Oncol. 2008 Feb 1;26(4):585-91. doi: 10.1200/JCO.2007.13.9881. Epub 2008 Jan 2. PMID 18172188
- [Background] Roach M 3RD, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D, Lawton C, Shipley W, Cox J. Predicting long-term survival, and the need for hormonal therapy: a meta-analysis of RTOG prostate cancer trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):617-27. doi: 10.1016/s0360-3016(00)00577-0. PMID 10837944